CLINICAL TRIAL: NCT00485628
Title: An Open-Label, Dose Titration Safety Study of Atomoxetine Hydrochloride in Outpatient Japanese Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Safety Study in Outpatient Japanese Children With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5286; B4Z-JE-LYBD
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride

SUMMARY:
Evaluate the safety and efficacy of atomoxetine in Japanese pediatric patients with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 6 - 18 years of age
* Patients must meet DSM-IV diagnostic criteria for ADHD
* Patient must be able to swallow capsules
* Patients must be of normal intelligence
* Laboratory results must show no significant abnormalities

Exclusion Criteria:

* Patients who weigh less than 15 kg or more than 75 kg at study entry
* Patients who have a documented history of bipolar disorder or any history of psychosis
* Patients taking any antipsychotic medication within 26 weeks of visit 1
* Patients with a severe history of allergies
* Patients taking methylphenidate

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2003-04; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to assess whether treatment with 1.8 mg/kg/day of atomoxetine will be safe and tolerable in a population of Japanese pediatric patients aged 6 through 18 years.

SECONDARY OUTCOMES:
To investigate the symptom scores in the ADHDRS-J at baseline and with atomoxetine therapy.
To evaluate the plasma concentration of atomoxetine, 4-hydroxyatomoxetine and N-desmethylatomoxetine

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo, Japan

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com